CLINICAL TRIAL: NCT06758037
Title: A Single-arm, Multicenter Phase II Clinical Study of HiR+X Therapy for Newly Diagnosed Diffuse Large B-cell Lymphoma (DLBCL) in Elderly Patients Intolerant to Chemotherapy, Guided by Molecular Subtyping and Clinical Characteristics.
Brief Title: Clinical Study of HiR+X Therapy for Newly Diagnosed Elderly Patients with DLBCL Intolerant to Chemotherapy
Acronym: HiR+X
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Lixia Sheng, Chief Physician, First Affiliated Hospital of Ningbo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-138A-02; 2024-138A-02 (Other: The Medical Ethics Committee of the First Affiliated Hospital of Ningbo University)
Record Dates: First submitted 2025-01-02; First posted 2025-01-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: DLBCL; Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; genetic subtypes; Zebtorizumab; Lenalidomide; unfit
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Drug Therapy; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with newly diagnosed, CD20+, elderly, chemotherapy-intolerant DLBCL (Experimental): All patients will receive one cycle of HiR (Zebtorizumab, Lenalidomide) induction therapy. On the first day of enrollment, tissue NGS and peripheral blood ctDNA will be submitted for testing. For the remaining six cycles, the added drug (X) will be determined based on the NGS molecular typing results. Please refer to the grouping scheme for details.
  HiR+X Dosing Scheme:
  Hi: Zebtorizumab 375mg/m², d1; R: Lenalidomide 10-25mg d1-10 (maximum tolerated dose)
  X:
  For MCD/BN2/TP53: Ocalivumab 150mg qd For EZB: Chidamide 30mg biw
  For N1-like and nonspecific types:
  If EBV-positive: PD-1 monoclonal antibody 200mg Q3W
  Interventions: Drug: Drug therapy

INTERVENTIONS:
Drug: Drug therapy — All patients will receive one cycle of HiR (Zebtorizumab, Lenalidomide) induction therapy. On the first day of enrollment, tissue NGS and peripheral blood ctDNA will be submitted for testing. For the remaining six cycles, the added drug (X) will be determined based on the NGS molecular typing results. Please refer to the grouping scheme for details.
  HiR+X Dosing Scheme:
  Hi: Zebtorizumab 375mg/m², d1; R: Lenalidomide 10-25mg d1-10 (maximum tolerated dose)
  X:
  For MCD/BN2/TP53: Ocalivumab 150mg qd For EZB: Chidamide 30mg biw
  For N1-like and nonspecific types:
  If EBV-positive: PD-1 monoclonal antibody 200mg Q3W
  Other Names: Ocalivumab; Chidamide; PD-1 monoclonal antibody

SUMMARY:
To explore the application of HiR (Zebtorizumab, Lenalidomide) + X (targeted drug) guided by NGS molecular typing, the aim is to assess the therapeutic efficacy and safety in newly diagnosed unfit or frail elderly patients with DLBCL aged ≥70 years, and to investigate the genetic subtypes that may benefit from HiR-X.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years;
2. ECOG score 0-3;
3. Rated as "unfit" or "frail" on the simplified geriatric assessment (sGA);
4. Histologically confirmed CD20-positive diffuse large B-cell lymphoma [diagnostic criteria according to WHO 2016], excluding transformed type 2 DLBCL;
5. Previously untreated, newly diagnosed patients;
6. Cardiac, hepatic, and renal function: creatinine < 2 times the upper limit of normal (ULN); ALT (alanine aminotransferase) / AST (aspartate aminotransferase) < 2.5 x ULN; total bilirubin < 2 x ULN;
7. At least one measurable lesion;
8. Intolerance to standard CHOP chemotherapy regimen or unwillingness to receive chemotherapy;
9. Sufficient understanding and voluntary signing of the informed consent form.

Exclusion Criteria:

1. Patients with central nervous system involvement at the onset of the disease;
2. Known human immunodeficiency virus (HIV) infection;
3. Pregnant or lactating women;
4. Other tumors requiring treatment;
5. Uncontrolled active infection;
6. Active hepatitis with HBV-DNA copy number unable to be controlled within 2000/mL despite antiviral treatment;
7. Individuals who cannot understand, comply with the study protocol, or sign the informed consent form.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) at the end of 6 cycles | Each cycle consists of 21 days, with a total of 6 cycles.
  Complete response rate (CR) at the end of 6 cycles

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poddubnaya IV, Alekseev SM, Kaplanov KD, Lukavetskyy LM, Rekhtman GB, Dolai TK, Attili VSS, Bermudez CD, Isaev AA, Chernyaeva EV, Ivanov RA. Proposed rituximab biosimilar BCD-020 versus reference rituximab for treatment of patients with indolent non-Hodgkin lymphomas: An international multicenter randomized trial. Hematol Oncol. 2020 Feb;38(1):67-73. doi: 10.1002/hon.2693. Epub 2020 Jan 13. PMID 31724191
- [Background] Shi Y, Song Y, Qin Y, Zhang Q, Han X, Hong X, Wang D, Li W, Zhang Y, Feng J, Yang J, Zhang H, Jin C, Yang Y, Hu J, Wang Z, Jin Z, Su H, Wang H, Yang H, Fu W, Zhang M, Zhang X, Chen Y, Ke X, Liu L, Yu D, Chen G, Wang X, Jin J, Sun T, Du X, Cheng Y, Yi P, Zhao X, Ma C, Cheng J, Chai K, Luk A, Liu E, Zhang X. A phase 3 study of rituximab biosimilar HLX01 in patients with diffuse large B-cell lymphoma. J Hematol Oncol. 2020 Apr 16;13(1):38. doi: 10.1186/s13045-020-00871-9. PMID 32299513